CLINICAL TRIAL: NCT04941534
Title: AMBulatory Fetal ECG Monitoring in High Risk Pregnancies
Brief Title: This Clinical Study Evaluates the Performance and Safety of Biorithm Research Kit Versus CTG in Prenatal Monitoring of Pregnant Participants.
Status: Completed | Type: Observational
Sponsor: Biorithm Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: AMBER
Record Dates: First submitted 2021-06-22; First posted 2021-06-28 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Pregnancy
Keywords: antepartum monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This clinical study will evaluate the safety and comparative performance of Biorithm Research Kit vs CTG (gold standard) in prenatal monitoring of pregnant participants.

DETAILED DESCRIPTION:
The Biorithm Research Kit system used in this study consists of femom fetal monitor (known as fetal monitor), a digital gateway and a cloud storage. It's intended for monitoring of maternal and fetal physiological parameters. It includes non-invasive fetal monitor or device, that monitors fetal heart rate (FHR), maternal heart rate (MHR), and uterine activity (UA) in the antepartum period.

ELIGIBILITY:
Inclusion Criteria:

* Have a singleton pregnancy
* Should be at and above 28 weeks of pregnancy
* Should have a valid indication for antenatal FHR monitoring as part of their pregnancy management, as per local hospital policy
* Able to speak English or have access to an interpreter and provide Informed Consent

Exclusion Criteria:

* Participants with an intellectual or mental impairment
* Participants with a known allergy or hypersensitivity to ECG gel electrodes
* Participants in pain, with contractions or in labour
* Known fetal cardiac or genetic abnormality
* Participant with a pacemaker

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Participants would be recruited at the Day Assessment Unit who require CTG monitoring and meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Fetal Heart Rate (FHR) | 60 minutes
  FHR agreement between Biorithm Research Kit and standard of care (CTG)
Maternal Heart Rate (MHR) | 60 minutes
  MHR agreement between Biorithm Research Kit and standard of care (CTG)

CONTACTS AND LOCATIONS:
Overall Officials: Baskaran Thilaganathan, Principal Investigator — St-George's University Hospital
Locations (1):
- St George's University Hospital, London, United Kingdom

REFERENCES:
- [Derived] Liu B, Marler E, Thilaganathan B, Bhide A. Ambulatory antenatal fetal electrocardiography in high-risk pregnancies (AMBER): protocol for a pilot prospective cohort study. BMJ Open. 2023 Apr 13;13(4):e062448. doi: 10.1136/bmjopen-2022-062448. PMID 37055213
- [Derived] Liu B, Thilaganathan B, Bhide A. Effectiveness of ambulatory non-invasive fetal electrocardiography: impact of maternal and fetal characteristics. Acta Obstet Gynecol Scand. 2023 May;102(5):577-584. doi: 10.1111/aogs.14543. Epub 2023 Mar 21. PMID 36944583